CLINICAL TRIAL: NCT07245589
Title: Development of Quantitative MRI Neuroimaging Protocols at High Fields (3 Tesla) and Ultra-high Fields (7 Tesla) for Clinical Evaluation: Application to Multiple Sclerosis
Brief Title: Evaluation of the Clinical Contribution of Quantitative MRI in Neuro-imaging
Acronym: NormaBRAIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: RCAPHM22_0366; ID-RCB 2025-A00346-43 (Other: ANSM)
Record Dates: First submitted 2025-10-02; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MS Patients (Experimental)
  Interventions: Other: 3T MRI; Other: 7T MRI; Other: Clinical examination of MS patients; Other: Neuropsychological testing of MS patients
- Healthy Volunteers (Sham Comparator)
  Interventions: Other: 3T MRI; Other: 7T MRI; Other: Quality of life questionnaires

INTERVENTIONS:
Other: 3T MRI — For this intervention, subjects will undergo a 3T MRI. The duration of an MRI session will not exceed 1h30
Other: 7T MRI — For this intervention, healthy subjects and patients will undergo a 7T MRI. The duration of an MRI session will not exceed 1h30
Other: Clinical examination of MS patients — During this interevention, patients will be submitted to 2 tests the EDSS and the MSFC scores, assessing for physical and cognitive disabilities in patients.
  Arms: MS Patients
Other: Neuropsychological testing of MS patients — This interventions consists in submitting MS patients to diverses neurpsychological tests assessing various parameters:
  CSCT (Computerized Speed Cognitive Test) for speed of information processing. PASAT (Paced Auditory Serial Addition Test) fo executive functions, working memory and attention CVLT (California Verbal Learning Test) for verbal episodic memory BVMTR (Brief Visual Memory Test) for visual episodic memory Fluences for mental flexibility, attention, lexical access "Test des commissions" for Ecological evaluation of executive functions
  Moreover, patients will fill out auto-questionnaires of quality of life including: a self-questionnaire of laterality (EDINBURGH), fatigue (MFIS), depression (BECK), anxiety (STAI1 and STAI2), quality of life (MUSIQOL), sleep quality (PITTSBURGH) and cognitive complaint (PDQ) will be collected for the volunteers.
  Arms: MS Patients
Other: Quality of life questionnaires — This intervention consists in the completion diverse questionnaire assessing the quelity of life of the subject. These questionnaires include: a self-questionnaire of laterality (EDINBURGH), fatigue (MFIS), depression (BECK), anxiety (STAI1 and STAI2), quality of life (MUSIQOL), sleep quality (PITTSBURGH) and cognitive complaint (PDQ) will be collected for the volunteers.
  The completion of the self-questionnaires will take about 30 minutes.
  Arms: Healthy Volunteers

SUMMARY:
This study aims to develop the use of a quantitative MRI (qMRI) approach in neuroimaging for MS patients.

To achieve this task the main goals of this study will be:

* to standardize and optimize qMRI protocols (acquisition time, sensitivity)
* to acquire ranges of normative values of qMRI parameters as a function of age and sex at high fields (3 Tesla) and ultra-high fields (UHF for ultra-high field, 7 Tesla)
* To develop integrated tools for image processing and the generation of normative models of the healthy brain normative values
* To assess the clinical feasibility and the multicenter validation of the multiparametric tools proposed in the case of application to MS.

ELIGIBILITY:
Inclusion Criteria:

* For healthy volunteers :

  * Male or female aged 20 to 50
  * Subject with no history of previous or concomitant neurological and psychiatric diseases at the time of inclusion
  * Subject without a history of traumatic brain injury
  * Subject with no vascular history (arterial hypertension, stroke) or concomitant at the time of its inclusion
  * Subject has no history of chronic drug and/or alcohol abuse
  * Subject having received information regarding the study and having signed an informed consent
  * Beneficiary or entitled person to a social security scheme
* For MS patients

  * Male or female aged 18 to 52
  * Patient diagnosed with MS according to the
  * criteria of McDonald 2017
  * Patient presenting a maximum EDSS of 6
  * Patient with MS for less than 10 years of evolution
  * Patient having received information regarding the study and having signed an informed consent
  * Patient beneficiary or entitled to a plan of social security

Exclusion Criteria:

* For healthy subjects :

  * Subject presenting a contraindication to performing an MRI: pacemaker, presence of metal implants, claustrophobia.
  * Subject unable to maintain a supine position for a prolonged period
  * Subject in a period of exclusion from another research protocol at the time of signing consent/non-opposition form
  * Subjects covered by articles L1121-5 to 1121-8 of the Public Health Code (minor patient, adult patient under guardianship or curatorship, patient deprived of liberty, pregnant or breastfeeding woman)
* For MS patients

  * Subject presenting a contraindication to performing an MRI: pacemaker, presence of metal implants, claustrophobia.
  * Subject unable to maintain a supine position for a prolonged period
  * Subject in a period of exclusion from another research protocol at the time of signing consent/non-opposition form
  * Subjects covered by articles L1121-5 to 1121-8 of the Public Health Code (minor patient, adult patient under guardianship or curatorship, patient deprived of liberty, pregnant or breastfeeding woman)

Ages: 18 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 272 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Assessing the feasibility of an accelerated 3T and 7T qMRI approach | Day 1
  Sensitivity per unit of acquisition time (signal-to-noise ratio, SNR), short-term inter-examination reproducibility (intra-individual repeatability), as well as the minimum acquisition duration
To estimate standard values of qMRI biomarkers | Day 1
  qMRI metrics calculated over region of interests defined in white and gray matter, mean and standard deviation of qMRI parameters
To estimate normative inter-examination reproducibility of qMRI biomarkers | During the first visit at Day 1 and during the second visit at day 60
  Inter-examination reproducibility (intra-individual repeatability)

SECONDARY OUTCOMES:
To evaluate external reproducibility using 10 healthy subjects | Day 1
  Comparing healthy volunteers quantitative parameters with standard values on the same age (average +/- 1.96 standard deviation)
To Evaluate the clinical contribution of quantitative MRI on a population of 100 MS patients | Day 1
  Difference between MRI acquired data values and standard values (step 2), clinical contribution compared to the usual assessment (qualitative analysis).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Gui de Chauliac, Montpellier, France

IPD SHARING:
Plan to Share IPD: No